CLINICAL TRIAL: NCT04933526
Title: The Efficacy and Safety of Switching to Flumatinib Versus Dasatinib After Imatinib-related Low-grade Adverse Events in Patients With Chronic Myeloid Leukemia in Chronic Phase: an Randomized Controlled Trial.
Brief Title: The Efficacy and Safety of Switching to Flumatinib Versus Dasatinib After Imatinib-related Low-grade Adverse Events in CML-CP Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210609
Record Dates: First submitted 2021-06-09; First posted 2021-06-21 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia in Chronic Phase
Keywords: Chronic Myeloid Leukemia in Chronic Phase; Imatinib; Flumatinib; Dasatinib
MeSH Terms: interventions — flumatinib; Dasatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flumatinib (Active Comparator): 600mg QD orally form 1 to 12 months
  Interventions: Drug: Flumatinib
- Dasatinib (Placebo Comparator): 100mg QD orally form 1 to 12 months
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Flumatinib — Flumatinib 600mg QD orally form 1 to 12 months
  Arms: Flumatinib
Drug: Dasatinib — Dasatinib 100mg QD orally form 1 to 12 months
  Arms: Dasatinib

SUMMARY:
The purpose of this study is to explore the efficacy and safety of switching to flumatinib versus dasatinib after imatinib-related low-grade adverse events in patients with chronic myeloid leukemia in chronic phase (CML-CP) in China. This is a post-marketing, interventional, double-arm, prospective, open-label, randomized controlled study in CML-CP patients in China. Patients will be recruited consecutively from the study sites during the enrollment period. The enrolled patients will be given flumatinib or dasatinib under the conditions of informed consent and frequent monitoring according to the clinical guideline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Diagnosis of CML-CP with Ph+;
* ECOG 0, 1, or 2;
* Patients with imatinib-related Low-grade Adverse Events for more than 12 months and AE lasting for at least 2 months, or relapsed at least 3 times in the past 12 months;
* Ability to provide written informed consent prior to any study related screening procedures being done

Exclusion Criteria:

* Previously documented T315I mutation;
* Previous treatment with any other tyrosine kinase inhibitor except for imatinib;
* Prior accelerated phase or blast phase CML;
* Loss of CHR or cytogenetic response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of (CTCAE grading scale) of imatinib related chronic low grade non hematologic Adverse Event after switch to treatment with flumatinib or dasatinib at 3 months. | 3 months

SECONDARY OUTCOMES:
Rate of a Major Molecular Response (MMR) after the switch to flumatinib or dasatinibin the therapy. | 12 months
Time to optimal imatinib-related adverse event improvement. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China